CLINICAL TRIAL: NCT05752409
Title: Comparison of Esketamine-Propofol and Fentanyl-Propofol on Haemodynamics in Elderly Patients
Brief Title: Comparison of Esketamine-Propofol and Fentanyl-Propofol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: esketamine-Propofol
Record Dates: First submitted 2023-01-28; First posted 2023-03-02 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-01

CONDITIONS: Hemodynamics
Keywords: esketamine; propofol; hemodynamic effects; elderly patients
MeSH Terms: interventions — Ketamine; Esketamine; Propofol; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Propofol + esketamin 0.5 (Experimental): 1mg•kg-1propofol, 0.5 mg•kg-1esketamin, 1 μg•kg-1 fentanyl and 0.15 mg•kg-1 cis-atracurium was administered intravenously in one minute.
  Interventions: Drug: The median dose of esketamine
- Propofol+ esketamin 0.75 (Experimental): 1mg•kg-1propofol, 0.75 mg•kg-1esketamin, 1 μg•kg-1 fentanyl and 0.15 mg•kg-1 cis-atracurium was administered intravenously in one minute.
  Interventions: Drug: The high dose of esketamine
- Propofol (Active Comparator): 2 mg•kg-1propofol, 1 μg•kg-1 fentanyl and 0.15 mg•kg-1 cis-atracurium was administered intravenously in one minute.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: The median dose of esketamine — 1mg•kg-1propofol and 0.5 mg•kg-1esketamine for general anesthesia induction.
  Other Names: s(+)ketamine
  Arms: Propofol + esketamin 0.5
Drug: The high dose of esketamine — 1mg•kg-1propofol and 0.75 mg•kg-1esketamine for general anesthesia induction.
  Other Names: s(+)ketamine
  Arms: Propofol+ esketamin 0.75
Drug: Propofol — 2mg•kg-1propofol for general anesthesia induction.
  Other Names: Propofol 10 mg/ml Injection
  Arms: Propofol

SUMMARY:
Propofol is widely used as an induction agent during general anesthesia. The prevalent induction dose may be associated with unacceptable cardiovascular instability, especially in elderly patients.The combination of ketamine and propofol has been shown to balance the cardiodepressant effects. Esketamine is dextrorotatory structure of ketamine but with stronger analgesic effects and fewer adverse events.However, there have been no previous published reports on the use of esketamine combined with propofol during induction. The main aim of this study was to investigate the haemodynamic effects of esketamine with propofol for the elderly during induction with LMA( laryngeal mask airway) insertion.

DETAILED DESCRIPTION:
Propofol is widely used as an induction agent during general anesthesia. The prevalent induction dose may be associated with unacceptable cardiovascular instability, especially in elderly patients. 1.7(0.6) mg.kg-1 adjusted dosed propofol demonstrated by a large multicenter cohort is suitable to advanced patients over aged 65.

Ketamine increases heart rate and arterial blood pressure by its activation of the sympathetic nervous system. When it is used with propofol for induction of general anesthesia, the cardiostimulating effects of ketamine balance the cardiodepressant effects of propofol. Esketamine is dextrorotatory structure of ketamine but with stronger analgesic effects and fewer adverse events. A previous study has shown that the use of ketamine before induction with propofol preserves haemodynamic stability during LMA insertion. However, there have been no previous published reports on the use of esketamine combined with propofol in elderly patients for induction.

The main aim of this study was to investigate the haemodynamic effects of esketamine with propofol during induction with LMA insertion. The secondary aim was to investigate whether the administration of esketamine in induction would delay the emergence of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* age 》60 years
* American Society of Anesthesiologists (ASA) class I or II

Exclusion Criteria:

* contraindications to esketamine, such as glaucoma and large vascular aneurysms
* poorly controlled or untreated hypertension (systolic/diastolic blood pressure over 180/100 mmHg at rest)
* severe cardiopulmonary
* mental illness.
* LMA insertion failed.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-10-08 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
systolic blood pressure (T0) | before induction of anesthesia (T0; baseline)
  systolic blood pressure (SBP)
systolic blood pressure (T1) | at the end of anaesthesia induction (T1)
  systolic blood pressure (SBP)
systolic blood pressure (T2) | at the time before LMA insertion (T2)
  systolic blood pressure (SBP)
systolic blood pressure (T3) | at the end of LMA insertion (T3)
  systolic blood pressure (SBP)
systolic blood pressure (T4) | 5min after LMA insertion (T4)
  systolic blood pressure (SBP)
systolic blood pressure (T5) | 10min after LMA insertion (T5)
  systolic blood pressure (SBP)
diastolic blood pressure (T0) | before induction of anesthesia (T0; baseline)
  diastolic blood pressure (DBP)
diastolic blood pressure (T1) | at the end of anaesthesia induction (T1)
  diastolic blood pressure (DBP)
diastolic blood pressure (T2) | at the time before LMA insertion (T2)
  diastolic blood pressure (DBP)
diastolic blood pressure (T3) | at the end of LMA insertion (T3)
  diastolic blood pressure (DBP)
diastolic blood pressure (T4) | 5min after LMA insertion (T4)
  diastolic blood pressure (DBP)
diastolic blood pressure (T5) | 10min after LMA insertion (T5)
  diastolic blood pressure (DBP)
mean arterial pressure (T0) | before induction of anesthesia (T0; baseline)
  mean arterial pressure (MAP)
mean arterial pressure (T1) | at the end of anaesthesia induction (T1)
  mean arterial pressure (MAP)
mean arterial pressure (T2) | at the time before LMA insertion (T2)
  mean arterial pressure (MAP)
mean arterial pressure (T3) | at the end of LMA insertion (T3)
  mean arterial pressure (MAP)
mean arterial pressure (T4) | 5min after LMA insertion(T4)
  mean arterial pressure (MAP)
mean arterial pressure (T5) | 10min after LMA insertion(T5)
  mean arterial pressure (MAP)
heart rate (T0) | before induction of anesthesia (T0; baseline)
  heart rate (HR))
heart rate (T1) | at the end of anesthesia induction (T1)
  heart rate (HR))
heart rate (T2) | at the time before LMA insertion (T2)
  heart rate (HR))
heart rate (T3) | at the end of LMA insertion (T3)
  heart rate (HR))
heart rate (T4) | 5min after LMA insertion(T4)
  heart rate (HR))
heart rate (T5) | 10min after LMA insertion(T5)
  heart rate (HR))
the occurrence of hypotension | during general anesthesia, about 15 min.
  hypotension is defined as systolic blood pressure decreased above 30% preanesthesia level or mean blood pressure<65 mmHg.

SECONDARY OUTCOMES:
Recovery time | from the time of completion of the procedure to the time of returning to the guard
  Recovery time was the time patients are extubated and acquire 10 scores by assessed with Modified Aldrete Score.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Tan, Principal Investigator — Anesthesiology Department of Affiliated Eye and ENT Hospital, Fudan University
Locations (1):
- Anesthesiology Department of Affiliated Eye and ENT Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li J, Wang Z, Wang A, Wang Z. Clinical effects of low-dose esketamine for anaesthesia induction in the elderly: A randomized controlled trial. J Clin Pharm Ther. 2022 Jun;47(6):759-766. doi: 10.1111/jcpt.13604. Epub 2022 Jan 11. PMID 35018643
- [Background] Yang H, Zhao Q, Chen HY, Liu W, Ding T, Yang B, Song JC. The median effective concentration of propofol with different doses of esketamine during gastrointestinal endoscopy in elderly patients: A randomized controlled trial. Br J Clin Pharmacol. 2022 Mar;88(3):1279-1287. doi: 10.1111/bcp.15072. Epub 2021 Oct 8. PMID 34496448
- [Background] Tu W, Yuan H, Zhang S, Lu F, Yin L, Chen C, Li J. Influence of anesthetic induction of propofol combined with esketamine on perioperative stress and inflammatory responses and postoperative cognition of elderly surgical patients. Am J Transl Res. 2021 Mar 15;13(3):1701-1709. eCollection 2021. PMID 33841692
- [Background] Zheng Y, Xu Y, Huang B, Mai Y, Zhang Y, Zhang Z. Effective dose of propofol combined with a low-dose esketamine for gastroscopy in elderly patients: A dose finding study using dixon's up-and-down method. Front Pharmacol. 2022 Sep 20;13:956392. doi: 10.3389/fphar.2022.956392. eCollection 2022. PMID 36204220
- [Background] Wei W, Zhang A, Liu L, Zheng X, Tang C, Zhou M, Gu Y, Yao Y. Effects of subanaesthetic S-ketamine on postoperative delirium and cognitive function in elderly patients undergoing non-cardiac thoracic surgery: a protocol for a randomised, double-blinded, placebo-controlled and positive-controlled, non-inferiority trial (SKED trial). BMJ Open. 2022 Aug 1;12(8):e061535. doi: 10.1136/bmjopen-2022-061535. PMID 35914911
- [Background] Brinck ECV, Maisniemi K, Kankare J, Tielinen L, Tarkkila P, Kontinen VK. Analgesic Effect of Intraoperative Intravenous S-Ketamine in Opioid-Naive Patients After Major Lumbar Fusion Surgery Is Temporary and Not Dose-Dependent: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial. Anesth Analg. 2021 Jan;132(1):69-79. doi: 10.1213/ANE.0000000000004729. PMID 32167978
- [Background] Xu Y, Zheng Y, Tang T, Chen L, Zhang Y, Zhang Z. The effectiveness of esketamine and propofol versus dezocine and propofol sedation during gastroscopy: A randomized controlled study. J Clin Pharm Ther. 2022 Sep;47(9):1402-1408. doi: 10.1111/jcpt.13678. Epub 2022 Apr 30. PMID 35488787